CLINICAL TRIAL: NCT03624062
Title: MER3101: MAS-1 Adjuvanted Antigen-specific Immunotherapeutic for Prevention and Treatment of Type 1 Diabetes
Acronym: MER3101
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); Nova Immunotherapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 15-1352
Record Dates: First submitted 2018-07-23; First posted 2018-08-09 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: New onset
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 33 ug IBC in 0.25 mL MAS-1 emulsion (Other): 7 participants to be randomized between placebo and MAS-1 adjuvanted insulin B-chain (2:5) with a 33 ug IBC dose in 0.25 mL MAS-1 emulsion
  Interventions: Drug: MAS-1 adjuvanted Insulin B-chain
- 109 ug IBC in 0.25 mL MAS-1 emulsion (Other): 7 participants to be randomized between placebo and MAS-1 adjuvanted insulin B-chain (2:5) with a 109 ug IBC dose in 0.25 mL MAS-1 emulsion
  Interventions: Drug: MAS-1 adjuvanted Insulin B-chain
- 327 ug IBC in 0.25 mL MAS-1 emulsion (Other): 7 participants to be randomized between placebo and MAS-1 adjuvanted insulin B-chain (2:5) with a 327 ug IBC dose in 0.25 mL MAS-1 emulsion
  Interventions: Drug: MAS-1 adjuvanted Insulin B-chain
- TBD ug IBC in 0.25 mL MAS-1 emulsion (Other): 7 participants to be randomized between placebo and MAS-1 adjuvanted insulin B-chain (2:5) with the optimal IBC dose selected from the first 3 groups (either 33 µg, or 109 µg, or 327 µg IBC) in 0.25 mL MAS-1 emulsion
  Interventions: Drug: MAS-1 adjuvanted Insulin B-chain

INTERVENTIONS:
Drug: MAS-1 adjuvanted Insulin B-chain — MER3101 (MAS-1 adjuvanted insulin B chain (IBC)), is a white, free-flowing 30:70 (w/w) water-in-oil (W/O) emulsion. MER3101 contains in the aqueous (disperse) phase 33, 109, or 327 µg per 0.25 mL dose of IBC (Drug Substance) and the oil (continuous) phase is comprised of MAS-1 oil vehicle.

SUMMARY:
The study is a randomized, double-masked, placebo-controlled, Phase 1 dose-escalation clinical trial. The objective of the trial is to determine if IBC adjuvanted with MAS-1 is safe and will favor tolerogenic pathways to restore immunologic balance and reverse type 1 diabetes (T1D) autoimmunity.

DETAILED DESCRIPTION:
The study is a four-arm (cohort), single center, randomized, double-masked, placebo-controlled, dose-escalation clinical trial. In this Phase I study, subjects (5 active MER3101 per arm plus 2 MAS-1 placebo) will be randomized to receive two intramuscular doses at days 0 and 28 of either MAS-1 placebo emulsion or MAS-1 adjuvanted IBC at 33, 109, and 327 µg IBC in 0.25 mL MAS-1 adjuvanted emulsion, followed by an additional arm to receive the optimal IBC dose selected from the first 3 arms in 0.25 mL MAS-1 emulsion. All groups will receive standard intensive diabetes treatment with insulin and dietary management.

The primary endpoint is assess the safety and tolerability of 3 doses of progressively higher IBC antigen doses of the vaccine, at 0.25 mL of MAS-1 adjuvant emulsion. In addition, to determine if the vaccine induces a shift towards protection shown by increased levels of IL-4, IL-5, IL-10 and TGF-b and regulatory changes in insulin-specific T and B cells using novel reagents to detect these unique populations of cells in treated subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 18 and 45 years of age who meet the ADA standard T1DM criteria and are positive for at least 1 islet cell autoantibody.
2. Type 1-diabetes mellitus diagnosed within the previous 2 years at time of screening
3. Must have stimulated C-peptide levels ≥ 0.2 pmol/ml measured during a mixed meal tolerance test (MMTT) conducted at least 21 days from diagnosis of diabetes and within one month (37 days) of randomization
4. At least one month from last immunization
5. Must be willing to comply with intensive diabetes management
6. If participant is female with reproductive potential, she must have a negative pregnancy test and be willing to avoid pregnancy during the treatment period until 2 months after the last study drug administration.
7. Willing to forgo routine clinical immunizations during the first 100 days after initial study drug administration (COVID-19 vaccination is permitted 60 days following initial study drug administration)
8. Subjects must have HbA1c levels under 9.5 to be enrolled in the study.
9. At least 30 days from receiving a single dose COVID-19 vaccine or at least 30 days from completing a multi-dose COVID-19 vaccine series.

Exclusion Criteria:

1. Be currently pregnant or lactating, or anticipate getting pregnant during the treatment period until 2 months after the last study drug administration.
2. Ongoing use of medications known to influence glucose tolerance
3. Require use of systemic immunosuppressant(s)
4. Any significant diabetes complications such as renal disease (proteinuria or elevated Cr) and diabetic retinopathy
5. Have a history of malignancies
6. Be currently using non-insulin pharmaceuticals to affect glycemic control
7. Have any acute or chronic complicating medical issues or abnormal clinical laboratory results that interfere with study conduct or cause increased risk including neurological abnormalities.
8. Inability or unwillingness to comply with the provisions of this protocol
9. Have an active infection or positive tuberculosis test result.
10. Have serologic evidence of current or past HIV, Hep B, or Hep C infection.
11. Have a known history of hypersensitivity or allergy reactions to squalane or squalene based adjuvants or other components of the study immunogen
12. Subjects with a history or evidence of chronic kidney disease (serum creatinine> 1.5mg/dL)
13. Subjects with a history of proliferative diabetic retinopathy that has not been treated with laser therapy
14. Subjects with a history of neuropathy, foot ulcers, amputations, or kidney disease
15. Males of reproductive potential who are unwilling to use acceptable birth control during the treatment period through 2 months after the last study drug administration, unless the female partner is postmenopausal or surgically sterile.
16. Have current, confirmed COVID-19 infection

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2025-12-04 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 43 months
  Number of participants with Treatment-Related Adverse Events, and the frequency of Adverse Events, as Assessed by CTCAE v4.0. The rates of severe hypoglycemic and adverse events will be computed (total number of events divided by total patient years of follow-up) and the rates compared using a Poisson regression model.
Immunologic Analysis | 43 months
  T cell assays looking for IL-4, IL-5, IL-10, IL-13, TGFβ production and shift towards Treg and iNKT cell population.

SECONDARY OUTCOMES:
Mean C-peptide AUC value | 43 months
  The area under the stimulated C-peptide curve (AUC) over the first 2 hours of a mixed meal glucose tolerance test. The AUC is computed using the trapezoidal rule that is a weighted sum of the C-peptide values over the 120 minutes.
HbA1c value | 43 months
  The mean HbA1c over all follow-up values will be compared between the control and placebo group using a normal errors longitudinal analysis.
Insulin Use | 43 months
  The mean insulin dose (units/kg) over all follow-up values will be compared between the control and placebo group using a normal errors longitudinal analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gottlieb, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No